CLINICAL TRIAL: NCT04823910
Title: Personalizing Docetaxel Dosing in Advanced Prostate Cancer
Acronym: PARTNER
Status: Completed | Type: Observational
Sponsor: Physiomics (Industry)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/41
Record Dates: First submitted 2021-03-23; First posted 2021-04-01 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with advanced prostate cancer are often treated with the chemotherapy drug docetaxel. The manufacturers of this drug suggest using the same dose of drug per m² body surface area for all patients. However we know that individuals end up with more or less of the drug circulating in their blood even after they have been given the same dose.

A software program (a "Dosing Tool") has been developed to provide information to doctors on how docetaxel will affect individual patients. The program may help doctors to make informed decisions about exactly how much drug to give to different people.

The purpose of the PARTNER study is to gather information from blood tests on patients being treated with docetaxel to help in the further development of the Dosing Tool. Some of these blood tests would have been taken anyway as part of patients' routine treatment. Others are extra for this study. Apart from the additional blood tests, everyone who enters the study is treated just as they would normally be if they were not taking part in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with metastatic prostate cancer (hormone sensitive or castrate resistant) and histologically confirmed
* Metastatic at disease onset or relapsed disease
* A treatment decision has been made to start a course of docetaxel as part of their standard of care treatment in accordance with the drug's label and the treating clinician's judgement
* Patient has not received a previous cycle of docetaxel within 8 weeks of the date of enrolment
* Life expectancy > 12 weeks
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

- Patients with autoimmune disease receiving active treatments Participant is unable to give informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient with metastatic prostate cancer due to start treatment with docetaxel
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Measured vs predicted absolute neutrophil count over time between weeks three and six of docetaxel treatment | The tool will be used to predict the level of neutropenia between the second and third doses of docetaxel (so between weeks three and six of treatment)

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, United Kingdom